CLINICAL TRIAL: NCT05890768
Title: The Relationship Between the Efficacy of Lumateperone and Central Glutamate and Dopaminergic Metabolism: A Comparison With Risperidone in First Episode Psychosis
Brief Title: Relationship Between Efficacy of Lumateperone and Brain Glutamate and Dopamine
Acronym: Lumafep
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: PI was unable to meet 1 year recruitment goal
Sponsor: University of New Mexico (Other)
Responsible Party: Principal Investigator, Juan R Bustillo, Professor of Psychiatry, University of New Mexico
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 22-396
Record Dates: First submitted 2023-02-22; First posted 2023-06-06 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-03

CONDITIONS: Psychosis
MeSH Terms: conditions — Psychotic Disorders | interventions — lumateperone; Risperidone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Lumateperone (Experimental): Lumateperone 42 mg capsule 1 PO QD for 6 weeks
  Interventions: Drug: Lumateperone
- Risperidone (Active Comparator): Risperidone starts 1 mg capsule PO QD for 1 week; then titrated blindly per clinical response and tolerability up to: 2 mg capsule QD starting in week 2; up to 3 mg capsule QD starting in week 3; and up to 4 mg capsule QD starting in week 4. Total risperidone exposure of 6 weeks.
  Interventions: Drug: Risperidone

INTERVENTIONS:
Drug: Lumateperone — FDA approved antipsychotic drug
  Other Names: Caplyta
  Arms: Lumateperone
Drug: Risperidone — FDA approved antipsychotic drug
  Other Names: Risperdol
  Arms: Risperidone

SUMMARY:
This study will examine the differential relationships between antipsychotic efficacy and changes in dopaminergic and glutamatergic brain metabolism in lumateperone and risperidone treated early psychosis patients. Baseline glutamate and dopamine brain scans, and symptom severity measures will be collected, followed by repeated measures at 6 weeks. Half of the early psychosis patients will be treated with lumateperone, half with risperidone. Healthy control subejcts will also be examined once.

DETAILED DESCRIPTION:
Efficacy. To examine the differential relationships between antipsychotic efficacy and changes in central dopaminergic and glutamatergic metabolism in lumateperone and risperidone treated early psychosis patients. Hypothesis 1a). Lumateperone efficacy will be directly related to both striatal neuromelanin and medial cingulate glutamate changes. Hypothesis 1b). With risperidone, the relationship with efficacy will be restricted to striatal neuromelanin changes. Brain glutamate and dopamine measures will be collected once in healthy controls to assist in the interpretation of baseline psychosis findings.

Safety. To examine the differential extra-pyramidal and peripheral metabolic side-effects in lumateperone and risperidone-treated early psychosis patients. Hypothesis 2a). Risperidone will cause more EPS than lumateperone, and this will be related to greater increases in prolactin. Hypothesis 2b). Risperidone will cause greater weight gain than lumateperone, and this will be related to increments in plasma lipids.

Background:

Lumateperone is an effective atypical antipsychotic with dopamine, serotonin and glutamate effects, a benign safety profile in terms of EPS and metabolic syndrome and the advantage of a single dose. Efficacy and safety have been established compared to placebo in chronically-ill psychotic patients. However, lumateperone has not been tested against an active comparator or examined in first episode psychosis. With the recognition of the importance of reducing duration of untreated psychosis, establishing efficacy and safety of antipsychotics early in psychosis becomes critical. Early psychosis patients tend to respond more robustly than chronically ill patients, but may be more sensitive to side-effects. In addition, because of the absent or minimal previous antipsychotic exposure, an early psychosis sample offers a better opportunity to examine brain mechanisms underlying efficacy of novel compounds.

Glutamate abnormalities have been documented in schizophrenia mainly with single-voxel proton magnetic resonance spectroscopy (1H-MRS). Whole brain measurement of glumate (glutamate plus glutamine i.e.: Glx) with three dimentional echo planar spectroscopic imaging (3D-EPSI) and magnatic resonance scanning of neuromelanin, a sensitive proxy for dopamine concentration in the substantia nigra (S-N) has been recently implemented. The S-N is the origin of the dorsal-striatal terminal fields, where an increased dopamine release has been documented in-vivo in schizophrenia and bipolar-I subjects with positron emission tomography (PET). The lumateperone effects on brain dopamine and glutamate have been documented in rodent models of psychosis. This pilot study is proposed to examine the in-vivo effects of lumateperone on central measures of dopamine and glutamate metabolism and their relationship with efficacy, in early psychosis patients.

Significance. There are three significant specific implications for this proposal. First, data supporting the efficacy and tolerability of lumaterperone in first episode psychosis will encourage clinical use of this agent early in the course of schizophrenia and other related disorders. The single dose profile of lumateperone is clearly an advantage in these patients who often have compliance issues. Second, identifying the location of glutamatergic deficits is critical to inform probe placement for future neuromodulation studies, aimed to improve persistent psychotic symptoms. For example, if a particular cortical area (like the medial cingulate) has persistently increased Glx in partially-responsive patients, low-frequency transcranial magnetic stimulation (TMS) targeting the medial cingulate may result in symptomatic improvement for patients who fail available antipsychotic therapy. Alternatively, clinically-relevant reductions in Glx would support high-frequency TMS targeting specific locations. Finally, these studies will also inform anatomical site selection for future postmortem studies of schizophrenia and bipolar-I aimed at examining the molecular underpinnings of these illnesses. This is critical for the development of novel compounds for psychosis that go beyond DA-2 blockade.

Experimental Design and Methods. Subjects. Two groups at baseline: first episode psychosis (FEP) patients and HVs. Subsequently, FEP will be randomized to risperidone or lumateperone for 6 weeks. All FEP subjects will be scanned twice with MRI for 3D 1H-MRS and S-N neuromelanin, at baseline and following 6 weeks of assigned antipsychotic therapy. The HV group will be scanned once at baseline.

Clinical phases of the study. The study will have three clinical phases: Screening, Double Blind and Transition.

i) Screening. After informed consent, subjects will be screened for inclusion and exclusion criteria. If included, subjects will complete a SCID interview and a medical history. HV will also complete the MATRICS cognitive battery, one MRI scan and will be finished with the study. FEP will complete baseline MRI and laboratory work (CBC, UA, chemistry, TSH, liver panel, prolactin, lipids and fasting blood sugar -FBS) as well as a physical exam.

ii) Double Blind. Baseline clinical measures will include psychopathology and movement disorder ratings. FEP will be randomized 1:1 at baseline to treatment with lumateperone (single dose 42 mg/day) vs. risperidone (1 mg tablet, target dose between 1 to 4 mg/day). Tablets will be blinded and a 1-week supply will be dispensed by the research pharmacy staff at each visit, following clinical assessments by the research psychiatrist. Patients will take between 1 and 4 tablets in the evening of blinded medication targeting psychotic/manic symptoms. The following un-blinded supplemental psychotropic medications will be allowed at the discretion of the treating psychiatrist: a) benztropine 1- 4 mg/day (for parkinsonism or dystonia); b) lorazepam 1-4 mg/day (for akathisia, anxiety or insomnia); c) propranolol 20-120 mg/day (for akathisia); and d) trazodone 50 to 200 mg/day for insomnia. These supplemental medicines will not be provided by the research pharmacy as part of the study. The subject will get a regular prescription to fill at his/her local pharmacy.

Patients will be seen weekly by the research psychiatrist and clinical coordinator to assess clinical response, tolerability, compliance and to adjust the blinded and any supplemental medication. The end of study (after 6 weeks of treatment) will also include the MATRICS, the second MRI and the second set of blood-work (prolactin, lipids and FBS).

If patients experience any significant persistent intolerance to the assigned treatment (e.g.: parkinsonism that does not improve with benztropine or akathisia despite treatment with propranolol or lorazepam), their initial medication will be blindly switched to the alternative anti-psychotic. If the blinded medication switch occurs at or after 3 weeks of treatment with the original drug, the end of study assessments will be advanced to be completed as close as possible to the date of switching medications. If the switching occurs before 3 weeks of treatment, the end of study assessments will take place as planned, after a total of 6 weeks of blinded treatment (the goal is to ensure the maximum length of exposure to a particular antipsychotic before end of study assessments are implemented). If the patient's psychotic/manic symptoms are not responding as expected, the blinded medication will be gradually increased (up to 4 tab per day). However, if lack of response persists, the research psychiatrist will also have the option to switch the medication blindly (because of the gradual titration, we expect the medication switch due to lack of response to be very rare). End of study assessments will be advanced as when switching due to intolerance.

iii) Transition Finally, patients will be transitioned to open-label antipsychotic treatment with lumateperone (provided by study sponsor for up to 6 months) or to any other agent as per standard of care (for which the patient will be responsible). Patients will be seen weekly for 4 weeks by the research psychiatrist for stabilization on the selected treatment before being referred back to a community-based provider of the patient's choosing. Any other therapies, pharmacological and psychosocial, that are consistent with the standard of care will also be recommended to the subject during this transition phase.

c). Magnetic Resonance. MR scans will be performed once at baseline for all subjects and once after 6 weeks of double-blind treatment for FEP. The protocol consists of structural MRI, Neuromelanin and EPSI scans.

d). Clinical Ratings. Patients will be evaluated for psychopathology with: the Positive And Negative Symptoms rating Scale (PANSS), mania with the Young Mania Rating Scale, depressive symptoms with the Calgary Depression Scale and the Columbia Suicide Severity Rating Scale. They will be assessed for movement side effects with the Simpson-Angus Scale (SAS) for parkinsonism, Barnes Akathisia Scale (BAS) and the Assessment of Involuntary Movement (AIMS) scale for tardive dyskinesia.

e). Neurocognitive and functional measures. The MATRICS, the standard in psychosis research, is an overall neurocognitive outcome and will be collected in all subjects once. The MATRICS evaluates several domains: processing speed, attention/vigilance, working memory, verbal learning, visual learning, reasoning & problem solving, and social cognition. It will be collected once at baseline in HV and once at the end of 6 weeks of treatment in FEP (so that it better reflects the underlying cognitive capacity apart from the impact of acute psychosis).

Functional outcome will be assessed at baseline with the Specific Levels of Functioning scale (SLOF). The SLOF is administered to the caregiver of a psychotic patient and examines 6 domains: personal care skills, physical functioning, interpersonal relationships, social acceptability, activities of community living and work skills. The Validation of Everyday Real-World Outcomes study found the SLOF to be most robustly related to performance-based indices of neurocognition and everyday living skills.

f). Laboratory measures. All FEP subjects will undergo baseline clinical measures to assess safety before starting double-blind treatment including hemogram (CBC), chemistry (chem7), hepatic function (hepatic panel), thyroid stimulating hormone (TSH) and urine analyses. To examine tolerability (as per Aim 2) serum prolactin, lipids and fasting blood sugar will be collected at baseline and following 6 weeks of double-blind treatment. All blood-work will be collected while fasting, in the AM. Also all subjects (FEP and HV) will have a urine drug screen done on the day of MR scanning. Finally, to prevent MRI exposure to pregnant females, a urine pregnancy test will be collected in all female participants of child-bearing age on the day of each MRI scans.

ELIGIBILITY:
Patient group:

* Inclusion:

  1. Diagnosis of DSM-5 schizophrenia, bipolar-I mania and mixed episodes with psychotic features, schizophreniform, schizoaffective, delusional, and unspecified schizophrenia spectrum and other psychotic disorders, established with SCID-P for DSM-5;
  2. age between 18 and 40 years old;
  3. antipsychotic exposure no greater than 50 mg of olanzapine equivalents (Gardner et al. AJP, 2010) in the 7 days previous to baseline assessments.
* Exclusion:

  1. neurological disorder, intellectual disability, history of severe head trauma (unconciousness >10 min);
  2. diagnosis of active substance use disorder (except for nicotine and cannabinoids [cannabinoids use is a risk factor for psychosis]).

Healthy Volunteers (HV) group:

* Inclusion:

  a) age between 18 and 40 years old.
* Exclusion:

  1. current or past psychiatric disorder (assessed with the SCID-NP; subjects with past history of anxiety or depressive disorders receiving no active treatment in the previous 12 months may be included);
  2. past or current diagnosis of neurological disorder, history of severe head trauma or diagnosis of active substance use disorder (except for nicotine or cannabinoids); and c) history of a psychotic disorder in first-degree relatives.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2023-05-11 (Actual); Primary Completion 2024-02-28 (Actual); Study Completion 2024-02-28 (Actual)

PRIMARY OUTCOMES:
Positive symptoms | 6 weeks
  Positive Scale, Negative Scale, and General Psychopathology Scale (PANSS) positive symptoms. Scale: min 1 to max 7; higher score is worse outcome.

SECONDARY OUTCOMES:
Extrapyramidal symptoms | 6 weeks
  Simpson-Angus Scale (SAS). Scale: min 1 to max 5; higher score is worse outcome.
Correlation between positive symptoms and brain glutamate | 6 weeks
  Positive Scale, Negative Scale, and General Psychopathology Scale (PANSS; Scale: min 1 to max 7; higher score is worse outcome.) and brain spectroscopy glutamate
Correlation between positive symptoms and brain dopamine | 6 weeks
  Positive Scale, Negative Scale, and General Psychopathology Scale (PANSS, Scale: min 1 to max 7; higher score is worse outcome.) and brain neuromelanin
Correlation between extrapyramidal symptoms and brain dopamine | 6 weeks
  Simpson-Angus Scale (SAS, Scale: min 1 to max 5; higher score is worse outcome.) and brain neuromelanin
Correlation between SAS and prolactin | 6 weeks
  Simpson-Angus Scale (SAS, Scale: min 1 to max 5; higher score is worse outcome.) and serum prolactin
Correlation between weight gain and lipids | 6 weeks
  Weight gain and changes in cholesterol and triglycerides
Correlation between weight gain and blood sugar | 6 weeks
  Weight gain and changes in fasting blood sugar
Correlation between circular RNAs and positive symptoms | 6 weeks
  Positive Scale, Negative Scale, and General Psychopathology Scale (PANSS, Scale: min 1 to max 7; higher score is worse outcome.) and circular RNAs in blood

CONTACTS AND LOCATIONS:
Overall Officials: Juan Bustillo, MD, Principal Investigator — UNM HSC
Locations (1):
- University of New Mexico, Albuquerque, New Mexico, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Correll CU, Davis RE, Weingart M, Saillard J, O'Gorman C, Kane JM, Lieberman JA, Tamminga CA, Mates S, Vanover KE. Efficacy and Safety of Lumateperone for Treatment of Schizophrenia: A Randomized Clinical Trial. JAMA Psychiatry. 2020 Apr 1;77(4):349-358. doi: 10.1001/jamapsychiatry.2019.4379. PMID 31913424
- [Background] Snyder GL, Vanover KE, Zhu H, Miller DB, O'Callaghan JP, Tomesch J, Li P, Zhang Q, Krishnan V, Hendrick JP, Nestler EJ, Davis RE, Wennogle LP, Mates S. Functional profile of a novel modulator of serotonin, dopamine, and glutamate neurotransmission. Psychopharmacology (Berl). 2015 Feb;232(3):605-21. doi: 10.1007/s00213-014-3704-1. Epub 2014 Aug 15. PMID 25120104
- [Background] Addington J, Van Mastrigt S, Addington D. Duration of untreated psychosis: impact on 2-year outcome. Psychol Med. 2004 Feb;34(2):277-84. doi: 10.1017/s0033291703001156. PMID 14982133
- [Background] Lally J, MacCabe JH. Antipsychotic medication in schizophrenia: a review. Br Med Bull. 2015 Jun;114(1):169-79. doi: 10.1093/bmb/ldv017. Epub 2015 May 8. PMID 25957394
- [Background] Merritt K, Egerton A, Kempton MJ, Taylor MJ, McGuire PK. Nature of Glutamate Alterations in Schizophrenia: A Meta-analysis of Proton Magnetic Resonance Spectroscopy Studies. JAMA Psychiatry. 2016 Jul 1;73(7):665-74. doi: 10.1001/jamapsychiatry.2016.0442. PMID 27304221
- [Background] Bustillo JR, Upston J, Mayer EG, Jones T, Maudsley AA, Gasparovic C, Tohen M, Lenroot R. Glutamatergic hypo-function in the left superior and middle temporal gyri in early schizophrenia: a data-driven three-dimensional proton spectroscopic imaging study. Neuropsychopharmacology. 2020 Oct;45(11):1851-1859. doi: 10.1038/s41386-020-0707-y. Epub 2020 May 13. PMID 32403117
- [Background] Cassidy CM, Zucca FA, Girgis RR, Baker SC, Weinstein JJ, Sharp ME, Bellei C, Valmadre A, Vanegas N, Kegeles LS, Brucato G, Kang UJ, Sulzer D, Zecca L, Abi-Dargham A, Horga G. Neuromelanin-sensitive MRI as a noninvasive proxy measure of dopamine function in the human brain. Proc Natl Acad Sci U S A. 2019 Mar 12;116(11):5108-5117. doi: 10.1073/pnas.1807983116. Epub 2019 Feb 22. PMID 30796187
- [Background] McCutcheon RA, Krystal JH, Howes OD. Dopamine and glutamate in schizophrenia: biology, symptoms and treatment. World Psychiatry. 2020 Feb;19(1):15-33. doi: 10.1002/wps.20693. PMID 31922684
- [Background] Wang AM, Pradhan S, Coughlin JM, Trivedi A, DuBois SL, Crawford JL, Sedlak TW, Nucifora FC Jr, Nestadt G, Nucifora LG, Schretlen DJ, Sawa A, Barker PB. Assessing Brain Metabolism With 7-T Proton Magnetic Resonance Spectroscopy in Patients With First-Episode Psychosis. JAMA Psychiatry. 2019 Mar 1;76(3):314-323. doi: 10.1001/jamapsychiatry.2018.3637. PMID 30624573
- [Background] Thompson PM, Jahanshad N, Ching CRK, Salminen LE, Thomopoulos SI, Bright J, Baune BT, Bertolin S, Bralten J, Bruin WB, Bulow R, Chen J, Chye Y, Dannlowski U, de Kovel CGF, Donohoe G, Eyler LT, Faraone SV, Favre P, Filippi CA, Frodl T, Garijo D, Gil Y, Grabe HJ, Grasby KL, Hajek T, Han LKM, Hatton SN, Hilbert K, Ho TC, Holleran L, Homuth G, Hosten N, Houenou J, Ivanov I, Jia T, Kelly S, Klein M, Kwon JS, Laansma MA, Leerssen J, Lueken U, Nunes A, Neill JO, Opel N, Piras F, Piras F, Postema MC, Pozzi E, Shatokhina N, Soriano-Mas C, Spalletta G, Sun D, Teumer A, Tilot AK, Tozzi L, van der Merwe C, Van Someren EJW, van Wingen GA, Volzke H, Walton E, Wang L, Winkler AM, Wittfeld K, Wright MJ, Yun JY, Zhang G, Zhang-James Y, Adhikari BM, Agartz I, Aghajani M, Aleman A, Althoff RR, Altmann A, Andreassen OA, Baron DA, Bartnik-Olson BL, Marie Bas-Hoogendam J, Baskin-Sommers AR, Bearden CE, Berner LA, Boedhoe PSW, Brouwer RM, Buitelaar JK, Caeyenberghs K, Cecil CAM, Cohen RA, Cole JH, Conrod PJ, De Brito SA, de Zwarte SMC, Dennis EL, Desrivieres S, Dima D, Ehrlich S, Esopenko C, Fairchild G, Fisher SE, Fouche JP, Francks C, Frangou S, Franke B, Garavan HP, Glahn DC, Groenewold NA, Gurholt TP, Gutman BA, Hahn T, Harding IH, Hernaus D, Hibar DP, Hillary FG, Hoogman M, Hulshoff Pol HE, Jalbrzikowski M, Karkashadze GA, Klapwijk ET, Knickmeyer RC, Kochunov P, Koerte IK, Kong XZ, Liew SL, Lin AP, Logue MW, Luders E, Macciardi F, Mackey S, Mayer AR, McDonald CR, McMahon AB, Medland SE, Modinos G, Morey RA, Mueller SC, Mukherjee P, Namazova-Baranova L, Nir TM, Olsen A, Paschou P, Pine DS, Pizzagalli F, Renteria ME, Rohrer JD, Samann PG, Schmaal L, Schumann G, Shiroishi MS, Sisodiya SM, Smit DJA, Sonderby IE, Stein DJ, Stein JL, Tahmasian M, Tate DF, Turner JA, van den Heuvel OA, van der Wee NJA, van der Werf YD, van Erp TGM, van Haren NEM, van Rooij D, van Velzen LS, Veer IM, Veltman DJ, Villalon-Reina JE, Walter H, Whelan CD, Wilde EA, Zarei M, Zelman V; ENIGMA Consortium. ENIGMA and global neuroscience: A decade of large-scale studies of the brain in health and disease across more than 40 countries. Transl Psychiatry. 2020 Mar 20;10(1):100. doi: 10.1038/s41398-020-0705-1. PMID 32198361
- [Background] Kapur S. Psychosis as a state of aberrant salience: a framework linking biology, phenomenology, and pharmacology in schizophrenia. Am J Psychiatry. 2003 Jan;160(1):13-23. doi: 10.1176/appi.ajp.160.1.13. PMID 12505794
- [Background] Wengler K, He X, Abi-Dargham A, Horga G. Reproducibility assessment of neuromelanin-sensitive magnetic resonance imaging protocols for region-of-interest and voxelwise analyses. Neuroimage. 2020 Mar;208:116457. doi: 10.1016/j.neuroimage.2019.116457. Epub 2019 Dec 11. PMID 31841683
- [Background] Cox RW. AFNI: software for analysis and visualization of functional magnetic resonance neuroimages. Comput Biomed Res. 1996 Jun;29(3):162-73. doi: 10.1006/cbmr.1996.0014. PMID 8812068
- [Background] Pauli WM, Nili AN, Tyszka JM. A high-resolution probabilistic in vivo atlas of human subcortical brain nuclei. Sci Data. 2018 Apr 17;5:180063. doi: 10.1038/sdata.2018.63. PMID 29664465
- [Background] Knudsen K, Fedorova TD, Hansen AK, Sommerauer M, Otto M, Svendsen KB, Nahimi A, Stokholm MG, Pavese N, Beier CP, Brooks DJ, Borghammer P. In-vivo staging of pathology in REM sleep behaviour disorder: a multimodality imaging case-control study. Lancet Neurol. 2018 Jul;17(7):618-628. doi: 10.1016/S1474-4422(18)30162-5. Epub 2018 Jun 1. PMID 29866443
- [Background] Javitt DC, Carter CS, Krystal JH, Kantrowitz JT, Girgis RR, Kegeles LS, Ragland JD, Maddock RJ, Lesh TA, Tanase C, Corlett PR, Rothman DL, Mason G, Qiu M, Robinson J, Potter WZ, Carlson M, Wall MM, Choo TH, Grinband J, Lieberman JA. Utility of Imaging-Based Biomarkers for Glutamate-Targeted Drug Development in Psychotic Disorders: A Randomized Clinical Trial. JAMA Psychiatry. 2018 Jan 1;75(1):11-19. doi: 10.1001/jamapsychiatry.2017.3572. PMID 29167877
- [Background] Gardner DM, Murphy AL, O'Donnell H, Centorrino F, Baldessarini RJ. International consensus study of antipsychotic dosing. Am J Psychiatry. 2010 Jun;167(6):686-93. doi: 10.1176/appi.ajp.2009.09060802. Epub 2010 Apr 1. PMID 20360319
- [Background] Verma G, Woo JH, Chawla S, Wang S, Sheriff S, Elman LB, McCluskey LF, Grossman M, Melhem ER, Maudsley AA, Poptani H. Whole-brain analysis of amyotrophic lateral sclerosis by using echo-planar spectroscopic imaging. Radiology. 2013 Jun;267(3):851-7. doi: 10.1148/radiol.13121148. Epub 2013 Jan 29. PMID 23360740
- [Background] Maudsley AA, Darkazanli A, Alger JR, Hall LO, Schuff N, Studholme C, Yu Y, Ebel A, Frew A, Goldgof D, Gu Y, Pagare R, Rousseau F, Sivasankaran K, Soher BJ, Weber P, Young K, Zhu X. Comprehensive processing, display and analysis for in vivo MR spectroscopic imaging. NMR Biomed. 2006 Jun;19(4):492-503. doi: 10.1002/nbm.1025. PMID 16763967
- [Background] Kay SR, Fiszbein A, Opler LA. The positive and negative syndrome scale (PANSS) for schizophrenia. Schizophr Bull. 1987;13(2):261-76. doi: 10.1093/schbul/13.2.261. PMID 3616518
- [Background] Young RC, Biggs JT, Ziegler VE, Meyer DA. A rating scale for mania: reliability, validity and sensitivity. Br J Psychiatry. 1978 Nov;133:429-35. doi: 10.1192/bjp.133.5.429. PMID 728692
- [Background] Addington D, Addington J, Maticka-Tyndale E. Assessing depression in schizophrenia: the Calgary Depression Scale. Br J Psychiatry Suppl. 1993 Dec;(22):39-44. PMID 8110442
- [Background] Bongiovi-Garcia ME, Merville J, Almeida MG, Burke A, Ellis S, Stanley BH, Posner K, Mann JJ, Oquendo MA. Comparison of clinical and research assessments of diagnosis, suicide attempt history and suicidal ideation in major depression. J Affect Disord. 2009 May;115(1-2):183-8. doi: 10.1016/j.jad.2008.07.026. Epub 2008 Sep 23. PMID 18814917
- [Background] Simpson GM, Angus JW. A rating scale for extrapyramidal side effects. Acta Psychiatr Scand Suppl. 1970;212:11-9. doi: 10.1111/j.1600-0447.1970.tb02066.x. No abstract available. PMID 4917967
- [Background] Barnes TR. A rating scale for drug-induced akathisia. Br J Psychiatry. 1989 May;154:672-6. doi: 10.1192/bjp.154.5.672. PMID 2574607
- [Background] Schooler NR, Kane JM. Research diagnoses for tardive dyskinesia. Arch Gen Psychiatry. 1982 Apr;39(4):486-7. doi: 10.1001/archpsyc.1982.04290040080014. No abstract available. PMID 6121550
- [Background] Nuechterlein KH, Green MF, Kern RS, Baade LE, Barch DM, Cohen JD, Essock S, Fenton WS, Frese FJ 3rd, Gold JM, Goldberg T, Heaton RK, Keefe RS, Kraemer H, Mesholam-Gately R, Seidman LJ, Stover E, Weinberger DR, Young AS, Zalcman S, Marder SR. The MATRICS Consensus Cognitive Battery, part 1: test selection, reliability, and validity. Am J Psychiatry. 2008 Feb;165(2):203-13. doi: 10.1176/appi.ajp.2007.07010042. Epub 2008 Jan 2. PMID 18172019
- [Background] Kern RS, Nuechterlein KH, Green MF, Baade LE, Fenton WS, Gold JM, Keefe RS, Mesholam-Gately R, Mintz J, Seidman LJ, Stover E, Marder SR. The MATRICS Consensus Cognitive Battery, part 2: co-norming and standardization. Am J Psychiatry. 2008 Feb;165(2):214-20. doi: 10.1176/appi.ajp.2007.07010043. Epub 2008 Jan 2. PMID 18172018
- [Background] Schneider LC, Struening EL. SLOF: a behavioral rating scale for assessing the mentally ill. Soc Work Res Abstr. 1983 Fall;19(3):9-21. doi: 10.1093/swra/19.3.9. PMID 10264257
- [Background] Harvey PD, Raykov T, Twamley EW, Vella L, Heaton RK, Patterson TL. Validating the measurement of real-world functional outcomes: phase I results of the VALERO study. Am J Psychiatry. 2011 Nov;168(11):1195-201. doi: 10.1176/appi.ajp.2011.10121723. Epub 2011 May 15. PMID 21572166
- [Background] Bustillo JR, Lauriello J, Rowland LM, Thomson LM, Petropoulos H, Hammond R, Hart B, Brooks WM. Longitudinal follow-up of neurochemical changes during the first year of antipsychotic treatment in schizophrenia patients with minimal previous medication exposure. Schizophr Res. 2002 Dec 1;58(2-3):313-21. doi: 10.1016/s0920-9964(02)00210-4. PMID 12409172
- [Background] Bustillo JR, Rowland LM, Mullins P, Jung R, Chen H, Qualls C, Hammond R, Brooks WM, Lauriello J. 1H-MRS at 4 tesla in minimally treated early schizophrenia. Mol Psychiatry. 2010 Jun;15(6):629-36. doi: 10.1038/mp.2009.121. Epub 2009 Nov 17. PMID 19918243

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-05-01): https://cdn.clinicaltrials.gov/large-docs/68/NCT05890768/Prot_SAP_000.pdf
  • Informed Consent Form (2023-05-01): https://cdn.clinicaltrials.gov/large-docs/68/NCT05890768/ICF_001.pdf